CLINICAL TRIAL: NCT07063017
Title: Comparative Effects of Post-isometric Relaxation and Active Release Technique in Pain, Range of Motion and Disability in Patients With Deep Gluteal Syndrome
Brief Title: Comparative Effects of Post-isometric Relaxation and Active Release Technique Patients With Deep Gluteal Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR &AHS/24/0161 Ujala
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Deep Gluteal Syndrome
Keywords: Pain; Disability; Range of motion
MeSH Terms: conditions — Hip socket neuropathy; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post- Isometric Relaxation (Experimental): Post Isometric Relaxation Technique to Piriformis; Lay the patient in the supine position and have the practitioner stand on the same side as the affected piriformis muscle. Bend the knee of the affected side and place the foot of that side on the lateral aspect of the opposite knee. Have the practitioner push knee medially until meeting the restrictive barrier. Have the patient push against the practitioner's resistance for 3 to 5 seconds, allow for a period of isometric relaxation, then engage a new barrier; repeat three times. Return the patient to a neutral position and reassess using supine or prone piriformis testing.
  Interventions: Other: Post- Isometric Relaxation
- Active Release Technique (Experimental): Active Release Technique:
  Patient position is side lying on the sound side. Therapist stands behind the patient. The upper leg must be in flexion on knee and slight extension Now apply pressure with both thumbs on piriformis and ask patient to flex and extend his hip and also external and internal rotation on hip in flexion. The gluteal muscle is taken from a shortened position to a fully lengthened position while the physiotherapist's contact hand holds tension longitudinally along the soft tissue fibers.
  Interventions: Other: Active Release Technique

INTERVENTIONS:
Other: Post- Isometric Relaxation — Post Isometric Relaxation Technique to Piriformis; Lay the patient in the supine position and have the practitioner stand on the same side as the affected piriformis muscle. Bend the knee of the affected side and place the foot of that side on the lateral aspect of the opposite knee. Have the practitioner push knee medially until meeting the restrictive barrier. Have the patient push against the practitioner's resistance for 3 to 5 seconds, allow for a period of isometric relaxation, then engage a new barrier; repeat three times. Return the patient to a neutral position and reassess using supine or prone piriformis testing.
  Arms: Post- Isometric Relaxation
Other: Active Release Technique — Patient position is side lying on the sound side. Therapist stands behind the patient. The upper leg must be in flexion on knee and slight extension Now apply pressure with both thumbs on piriformis and ask patient to flex and extend his hip and also external and internal rotation on hip in flexion. The gluteal muscle is taken from a shortened position to a fully lengthened position while the physiotherapist's contact hand holds tension longitudinally along the soft tissue fibers.
  Arms: Active Release Technique

SUMMARY:
Deep gluteal syndrome included piriformis syndrome. Tight piriformis muscle gives symptoms of Sciatica in patients with Deep Gluteal Syndrome. Two different techniques which will be used to improve deep gluteal syndrome are Active release technique and Post-isometric relaxation. Active release therapy is a set of techniques for treating musculoskeletal problems. After feeling for the precise location of musculoskeletal dysfunction, practitioners aim to release affected tissues. The post-isometric relaxation technique begins by placing the muscle in a stretched position. Then an isometric contraction is exerted against minimal resistance. Relaxation and then gentle stretch follow as the muscle releases.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial and will be conducted in Riphah Rehabilitation Clinic Lahore. Non-probability consecutive sampling will be used to collect the data. Sample size of 46 subjects with age group between 35-55 years of both male and female will be taken. Data will be collected from the patients having present complaint of pain in buttock, low back and radiating to leg. Outcome measures will be taken using Numeric Pain Rating Scale (NPRS) for pain, Low Extremity Functional Scale for disability and Universal Goniometer (GU) for Range of Motion. An informed consent will be taken. Subjects will be selected on the basis of inclusion and exclusion criteria and will be equally divided into two groups by random number generator table. Both the Groups will receive hot pack, TENS and ultrasound as well as stretching exercises of piriformis while Group A will receive Post-isometric relaxation and Group B will receive Active release technique. Outcome measures will be measured at baseline and after 4 weeks. Data analysis will be done by SPSS version 21.

ELIGIBILITY:
Inclusion Criteria:

* •Age group between 35 and 55 years

  * Both gender male and female
  * Having pain and tenderness in gluteal space
  * Gluteal pain radiating through the posterior of thigh and lower limb

Exclusion Criteria:

* • Pregnancy

  * Malignancies
  * Degenerative spine disorders like lumber spondylosis, canal stenosis, spondylolisthesis, neural compressions due to intervertebral disc lesions
  * Any vertebral or hip fracture.
  * History of spinal surgery, TB spine, osteoarthritis, rheumatoid disease

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) | upto 4 weeks
  Patient level of pain will be assessed using this scale. This scale ranges from 0 to 10. 0 indicates "no pain" and 10 indicated "worst pain".
Universal Goniometer (UG) | upto 4 weeks
  The range of motion will be measured using universal goniometer. A universal goniometer has 3 parts, which include the following: A body is designed like a protractor and may form a full or half-circle. It has a scale for the measurement of the angle. The scale can extend from 0 to 180 degrees for half-circle models or 0 to 360 degrees for full-circle models.
Lower Extremity Functional Scale (LEFS) | upto 4 weeks
  The Lower Extremity Functional Scale (LEFS) is a questionnaire containing 20 questions about a person's ability to perform everyday tasks. The LEFS can be used by clinicians as a measure of patients' initial function, ongoing progress and outcome, as well as to set functional goals.

CONTACTS AND LOCATIONS:
Overall Officials: Samrood Akram, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Ittefaq Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kizaki K, Uchida S, Shanmugaraj A, Aquino CC, Duong A, Simunovic N, Martin HD, Ayeni OR. Deep gluteal syndrome is defined as a non-discogenic sciatic nerve disorder with entrapment in the deep gluteal space: a systematic review. Knee Surg Sports Traumatol Arthrosc. 2020 Oct;28(10):3354-3364. doi: 10.1007/s00167-020-05966-x. Epub 2020 Apr 3. PMID 32246173
- [Background] Hernando MF, Cerezal L, Perez-Carro L, Abascal F, Canga A. Deep gluteal syndrome: anatomy, imaging, and management of sciatic nerve entrapments in the subgluteal space. Skeletal Radiol. 2015 Jul;44(7):919-34. doi: 10.1007/s00256-015-2124-6. Epub 2015 Mar 5. PMID 25739706
- [Background] Naz S, Sheikh SA, Sulaman M, Abid S, Saeed E, Faraz K. EFFECTS OF ACTIVE RELEASE TECHNIQUE VERSUS MULLIGAN TECHNIQUE ON PAIN AND FUNCTIONAL DISABILITY IN PATIENT WITH DEEP GLUTEAL SYNDROME.
- [Background] Park JW, Lee YK, Lee YJ, Shin S, Kang Y, Koo KH. Deep gluteal syndrome as a cause of posterior hip pain and sciatica-like pain. Bone Joint J. 2020 May;102-B(5):556-567. doi: 10.1302/0301-620X.102B5.BJJ-2019-1212.R1. PMID 32349600
- [Background] Boyajian-O'Neill LA, McClain RL, Coleman MK, Thomas PP. Diagnosis and management of piriformis syndrome: an osteopathic approach. J Am Osteopath Assoc. 2008 Nov;108(11):657-64. doi: 10.7556/jaoa.2008.108.11.657. PMID 19011229
- [Background] Kage V, Ratnam R. Immediate effect of active release technique versus mulligan bent leg raise in subjects with hamstring tightness: a randomized clinical trial. Int J Physiother Res. 2014;2(1):301-4.
- [Background] Michel F, Decavel P, Toussirot E, Tatu L, Aleton E, Monnier G, Garbuio P, Parratte B. The piriformis muscle syndrome: an exploration of anatomical context, pathophysiological hypotheses and diagnostic criteria. Ann Phys Rehabil Med. 2013 May;56(4):300-11. doi: 10.1016/j.rehab.2013.03.006. Epub 2013 Apr 30. PMID 23684469
- [Background] Dworkin RH, O'Connor AB, Backonja M, Farrar JT, Finnerup NB, Jensen TS, Kalso EA, Loeser JD, Miaskowski C, Nurmikko TJ, Portenoy RK, Rice ASC, Stacey BR, Treede RD, Turk DC, Wallace MS. Pharmacologic management of neuropathic pain: evidence-based recommendations. Pain. 2007 Dec 5;132(3):237-251. doi: 10.1016/j.pain.2007.08.033. Epub 2007 Oct 24. PMID 17920770